CLINICAL TRIAL: NCT03533439
Title: Regional Haemoglobin Oxygen Saturation in the Splanchnic Circulation in Neonates With Gastroschisis; Quantifying and Qualifying the Role for Routine Monitoring
Brief Title: Regional Blood Saturation Levels in Gastroschisis
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2013/0117
Record Dates: First submitted 2018-04-23; First posted 2018-05-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2018-01

CONDITIONS: Gastroschisis; Intestinal Ischemia
MeSH Terms: conditions — Gastroschisis | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Near infrared spectroscopy — Four channel measurement of regional haemoglobin oxygen saturation (SO2) in the blood of the bowel, kidney and brain of neonates with gastroschisis during reduction within a silo and after surgery will be performed.• Routine surgical procedure will be followed (clinically indicated silo placement and closure as is currently practised). There will be no change in the clinical practice in place during this pilot study. Clinical management will be as already practiced with the supervision of the consultant with clinical responsibility dictating management
  Other Names: in-vivo optical spectroscopy oximeter; INVOS (Somanetics, Troy, Mich).

SUMMARY:
Gastroschisis is one of the most common neonatal surgical conditions, and is increasing in incidence. Postnatal bowel ischemia leading to necrosis, bowel loss and short-bowel syndrome, occurs in a few instances, with significant impact. Intestinal gangrene occurs in up to 37%. The cause of the gangrene can be multifactorial. Contributing factors can be volvulus; venous engorgement with ensuing arterial compromise; constriction of the gut mesentery at the defect; and contribution of the hydrostatic effect of the column of bowel within a silo.

Theoretically, the increased hydrostatic pressure incurred by the bowel in a preformed silo, may decrease blood flow to the apex of the bowel and contribute to ischemia. However, this does not seem to be the norm, as most cases do well in the silo. Cases of intestinal ischaemia within the silo have been described in patients. Any objective measure of bowel perfusion and therefore viability which can aid clinical assessment and management may benefit patient outcome.

Near-infrared spectroscopy (NIRS) is used to noninvasively measure and monitor changes in the approximate regional haemoglobin oxygen saturation (SO2) in the blood. Measurement of oxygen saturation using NIRS is already in clinical application in other neonatal and paediatric medical and surgical diseases. NIRS has been recommended as a good trend indicator of changes in neonatal tissues oxygenation. NIRS-measured duration of cerebral oxygen desaturation is an accurate predictor of postoperative neurological injury in children undergoing cardiac surgery.

The investigators propose to use NIRS to measure SO2 in the intestinal bed in patients with gastroschisis and to ascertain if there is any clinical advantage to routine monitoring in these patients.

The aim of the study will be to:

1. Measure Gastrointestinal SO2 (GSO2) of the bowel within the silo of gastroschisis patients
2. Identify the clinical progress of patients with gastroschisis in the postnatal period
3. Identify any association of the measured GSO2 with the clinical outcome and any gastrointestinal complications

ELIGIBILITY:
Inclusion Criteria:

* Gastroschisis diagnosed antenatally or at birth

Exclusion Criteria:

* Associated congenital condition affecting respiratory system , cardiovascular system or global development
* Generalised sepsis

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn babies at neonatal unit
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
The incidence of intestinal ischemia requiring intervention and its correlation to measured GSO2 | Through study completion, an average of 6 weeks

SECONDARY OUTCOMES:
Time to full feeds | Through study completion, an average of 6 weeks
Changes in renal oxygenation measured by near infra-red spectroscopy | Through study completion, an average of 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Merrill McHoney, PhD, Principal Investigator — NHS Lothian

IPD SHARING:
Plan to Share IPD: Undecided